CLINICAL TRIAL: NCT02179242
Title: Randomized, Single Center Study to Determine if a Cardiac Rehabilitation Program Immediately Following Hospitalization Reduces Hospital Readmissions and Improves Quality of Life Outcomes in Heart Failure Patients.
Brief Title: Study to Evaluate the Effectiveness of Cardiac Rehabilitation (Rehab) for Acute Decompensated Heart Failure Patients on 6 Minute Walk Test and Quality of Life
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lower than expected accrual
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SH Cardiac Rehab for HF
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: cardiac rehab; heart failure; KCCQ; 6 minute walk test; readmission
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (No Intervention): This arm will receive routine care following their heart failure which includes no cardiac rehab intervention.
- Cardiac rehab (Experimental): This arm will receive cardiac rehab intervention 3 times per week for 4 weeks following discharge.
  Interventions: Other: Cardiac rehab

INTERVENTIONS:
Other: Cardiac rehab
  Arms: Cardiac rehab

SUMMARY:
The aim of the investigators' project is to determine if patients admitted with a primary diagnosis of heart failure to Sanford Health facilities in regional southeastern South Dakota demonstrate benefits in improvement in functional capacity, quality of life, and a reduction in hospital readmission rates from a cardiac rehab program immediately following a discharge for an acute decompensated heart failure diagnosis related inpatient hospitalization encounter. The investigators hypothesize that those that receive cardiac rehab will have improved quality of life and reduced readmission rates at 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Admitted with acute, decompensated heart failure
* Signed informed consent

Exclusion Criteria:

* Approved by Center for Medicare and Medicaid Services (CMS) to enroll in cardiac rehab
* Have an elective procedure that would interrupt their exercise program
* Unable to partake in an exercise program due to physical incapacities
* Pregnancy
* Unable to read and understand the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | 30 days
  Assess increased functional capacity, determined by the 6 minute walk test in the cardiac rehabilitation group compared to the routine care group at 4 weeks following hospital discharge

SECONDARY OUTCOMES:
Readmission | 30 days
  Determine if 30-day readmission rates are lower with those receiving cardiac rehabilitation compared to those receiving routine care
Readmission | 90 days
  Determine if 90-day readmission rates are lower with those receiving cardiac rehabilitation compared to those receiving routine care
KCCQ | 30 days
  Assess if those receiving cardiac rehabilitation have improved quality of life using the Kansas City Cardiomyopathy Questionnaire (KCCQ) classifications at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Orvar Jonsson, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Heart Hospital, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Davidson PM, Cockburn J, Newton PJ, Webster JK, Betihavas V, Howes L, Owensby DO. Can a heart failure-specific cardiac rehabilitation program decrease hospitalizations and improve outcomes in high-risk patients? Eur J Cardiovasc Prev Rehabil. 2010 Aug;17(4):393-402. doi: 10.1097/HJR.0b013e328334ea56. PMID 20498608
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):e6-e245. doi: 10.1161/CIR.0b013e31828124ad. Epub 2012 Dec 12. No abstract available. PMID 23239837
- [Background] Guazzi M, Dickstein K, Vicenzi M, Arena R. Six-minute walk test and cardiopulmonary exercise testing in patients with chronic heart failure: a comparative analysis on clinical and prognostic insights. Circ Heart Fail. 2009 Nov;2(6):549-55. doi: 10.1161/CIRCHEARTFAILURE.109.881326. Epub 2009 Sep 28. PMID 19919979
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Joseph SM, Novak E, Arnold SV, Jones PG, Khattak H, Platts AE, Davila-Roman VG, Mann DL, Spertus JA. Comparable performance of the Kansas City Cardiomyopathy Questionnaire in patients with heart failure with preserved and reduced ejection fraction. Circ Heart Fail. 2013 Nov;6(6):1139-46. doi: 10.1161/CIRCHEARTFAILURE.113.000359. Epub 2013 Oct 15. PMID 24130003
- [Background] Sauser K, Spertus JA, Pierchala L, Davis E, Pang PS. Quality of life assessment for acute heart failure patients from emergency department presentation through 30 days after discharge: a pilot study with the Kansas City Cardiomyopathy Questionnaire. J Card Fail. 2014 Jan;20(1):18-22. doi: 10.1016/j.cardfail.2013.11.010. Epub 2013 Dec 1. PMID 24296380
- [Background] Setoguchi S, Stevenson LW, Schneeweiss S. Repeated hospitalizations predict mortality in the community population with heart failure. Am Heart J. 2007 Aug;154(2):260-6. doi: 10.1016/j.ahj.2007.01.041. PMID 17643574